CLINICAL TRIAL: NCT00933738
Title: Evaluation of the Accuracy of the INRatio Prothrombin Time (PT) Monitoring System With a New Test Strip for the Oral Anticoagulation Therapy Patient in the Presence of Heparin and Low Molecular Weight Heparin (e.g., Enoxaparin or Dalteparin)
Acronym: ECLIPSE 03
Status: Completed | Type: Observational
Sponsor: Abbott RDx Cardiometabolic (Other)
Responsible Party: Keith Gran / Sr. Clinical Trial Manager, Biosite, Incorporated a subsidiary of Inverness Medical Innovations
Other Study IDs: BSTE-0120.a
Record Dates: First submitted 2009-07-03; First posted 2009-07-07 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Coagulation
Keywords: Patients needing OAT (Oral Anticoagulation Therapy)
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples to be retained for reference testing and banking.
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a multi-center study designed to evaluate the heparin insensitivity of the INRatio Prothrombin Time (PT) Monitoring System, utilizing an INRatio test strip additionally modified for low sample volume. The INRatio test strip is used for the quantitative determination of PT and International Normalized Ratio (INR) results in fingerstick blood from subjects on oral anticoagulation therapy (OAT) with warfarin. This study is designed to evaluate the accuracy of the modified INRatio test strip during heparin-warfarin bridge therapy with unfractionated heparin (UH) or low molecular weight heparin (LMWH), such as enoxaparin or dalteparin. These INR results will be compared to the INR results obtained on plasma from the same subjects as analyzed at a central laboratory with the heparin-insensitive reference method: the Sysmex CA-560 System. The levels of UH or LMWH in the plasma samples will be assessed using activated partial thromboplastin time (aPTT) and anti-factor-Xa assays respectively.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years of age or older).
* Willing and able to provide written informed consent and comply with study procedures.
* Receiving warfarin/heparin bridge therapy.
* Therapy with both warfarin and one of the heparins listed below must have been initiated for at least 12 hours before the first study specimens are obtained.
* UH (last known aPTT prior to enrollment (if available†) must confirm heparin has been administered)
* Dalteparin (last known anti-factor Xa prior to enrollment (if available†) must confirm heparin has been administered)
* Enoxaparin (last known anti-factor Xa prior to enrollment (if available†) must confirm heparin has been administered) † If a pre-study aPTT or anti-factor Xa is not available, subsequent testing of the study phlebotomy or a phlebotomy as a part of routine medical care taken before or during the time of the study phlebotomy must confirm the presence of heparin (unfractionated or low molecular weight) in order for that data point to be included in the analysis.

Exclusion Criteria

* Known or suspected hematocrit less than 25 or greater than 55%;
* Auto-immune disorders known to interfere with INR measurements, such as lupus or anti-phospholipid syndrome (APS)
* Already participated in this specific study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heparin bridging onto OAT with warfarin.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Loma Linda VA, Loma Linda, California
  - University of Colorado-Denver, Aurora, Colorado
  - Henry Ford Hospital, Detroit, Michigan
  - Emergency Medicine Research Group, Lansing, Michigan
  - Cardiac and Vascular Research Center of Northern Michigan, Petoskey, Michigan
  - International Heart Institute of Montana, Missoula, Montana
  - University of New Mexico, Albuquerque, New Mexico
  - New York Methodist Hospital, Brooklyn, New York
  - John T Mather Memorial Hospital, Port Jefferson, New York
  - Northwest Heart Center, Tomball, Texas
  - Swedish Medical Center, Seattle, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington